CLINICAL TRIAL: NCT04413279
Title: Intracanalicular Dexamethasone Used in Conjunction With LipiFlow for the Treatment of Meibomian Gland Dysfunction in Patients With Evaporative Dry Eye Disease and Evidence of Clinically Significant Inflammation
Brief Title: Lipiflow Treatment Alone vs. Lipiflow + Dextenza Treatment for Dry Eye Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eye Surgeons of Indiana (Network)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: The DIERKER Study
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lipiflow Only Group (Active Comparator): Patients with dry eye disease Lipiflow only
  Interventions: Procedure: LipiFlow Thermal Pulsation
- Lipiflow + Dextenza Group (Experimental): Patients with dry eye disease Lipiflow + Dextenza
  Interventions: Drug: Dexamethasone Intracanalicular Insert, 0.4mg with LipiFlow Thermal Pulsation

INTERVENTIONS:
Procedure: LipiFlow Thermal Pulsation — To manage patients with dry eye disease secondary to MGD
  Arms: Lipiflow Only Group
Drug: Dexamethasone Intracanalicular Insert, 0.4mg with LipiFlow Thermal Pulsation — to investigate the benefit of managing patients with DED secondary to MGD with a sustained release intracanalicular dexamethasone (0.4 mg) insert in addition to LipiFlow Thermal Pulsation
  Other Names: Dextenza
  Arms: Lipiflow + Dextenza Group

SUMMARY:
To evaluate the benefit of treatment with a physician administered intracanalicular dexamethasone insert in evaporative dry eye disease (DED) patients with meibomian gland disfunction (MGD) and underlying inflammation undergoing LipiFlow Thermal Pulsation.

DETAILED DESCRIPTION:
This prospective, open-label, single-center, non-randomized, investigator-sponsored clinical study seeks to investigate the benefit of managing patients with DED secondary to MGD with a sustained release intracanalicular dexamethasone (0.4 mg) insert in addition to LipiFlow Thermal Pulsation compared to LipiFlow Thermal Pulsation alone. In addition, this study will evaluate the ease of Dextenza insertion and the patient preference for therapy.

After screening a given patient for inclusion and exclusion criteria, and gaining informed consent, each eye will undergo LipiFlow Thermal Pulsation on the same day. The most symptomatic eye will be selected to receive DEXTENZA® insertion on the day of the procedure (study eye), while the other eye will be assigned to a receive a sham punctum dilation (control eye). If there is no obvious symptomatic difference, the right eye will receive the intracanalicular insert. Per patient, the study period will last for approximately 12 weeks after the LipiFlow procedure, consisting of one screening visit, one treatment v4isit and 3 post-procedure follow-up visits (week 1, week 4 and week 12). At week 1, week 4 and week 12, primary and secondary endpoints will be assessed alongside standard-of-care procedures. Adjusting for enrollment period, the study will last a total of approximately 4 months.

ELIGIBILITY:
Inclusion Criteria:

A patient's study eye must meet the following criteria to be eligible for inclusion in the study:

* 18 years of age or older
* Evaporative DED with MGD and clinically significant inflammation
* Willing and able to comply with clinic visits and study related procedures
* Willing and able to sign the informed consent form

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from the study:

* Patients under the age of 18.
* Pregnancy (must be ruled out in women of child-bearing age with pregnancy test)
* Active infectious systemic disease
* Active infectious ocular or extraocular disease
* Altered nasolacrimal flow of either acquired, induced, or congenital origin
* Hypersensitivity to dexamethasone
* Patient being treated with either topical, oral, or intravenous steroids
* Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in meibomian gland scores (expressibility and quality) | Assessed at Baseline, Week 1, Week 4 and Week 12
  As measured on a grading scale 1 to 4 and graded by the physician
Patient preference for | Assessed at Week 12
  As measured by COMTOL Survey

SECONDARY OUTCOMES:
Mean change in MMP-9 | Assessed at Baseline, Week 1, Week 4 and Week 12 Visit
  As measured by InflammaDry
Mean change in ocular surface staining | Assessed at Baseline, Week 1, Week 4 and Week 12 Visit
  As measured by sodium fluorescein and lissamine green
Mean change in tear break-up time (TBUT) | Assessed at Baseline, Week 1, Week 4 and Week 12 Visit
  As measured by TBUT testing
Mean change in tear osmolarity | Assessed at Baseline, Week 1, Week 4 and Week 12 Visit
  As measured by TearLab
Mean change in DEQ-5 | Assessed at Baseline, Week 1, Week 4 and Week 12 Visit
  As measured by DEQ-5 Questionnaire (Dry Eye Questionnaire. The DEQ-5 is comprised of 5 items: frequency of watery eyes, discomfort, and dryness (0-4 scale) and late day discomfort and dryness intensity (0-5 scale). Higher numbers indicate more severe symptoms.
Mean change in Best-corrected Visual Acuity (BCVA) | Assessed at Baseline, Week 1, Week 4 and Week 12 Visit
  As measured by ETDRS chart

CONTACTS AND LOCATIONS:
Overall Officials: Damon Dierker, OD, FAAO, Principal Investigator — Eye Surgeons of Indiana
Locations (1):
- Eye Surgeons of Indiana, Indianapolis, Indiana, United States